CLINICAL TRIAL: NCT06097884
Title: Healthy School mEAls With Less Salt：an Action to Reduce Salt Intake in School Meals for Children in Rural China（HEALS-child）
Brief Title: Healthy School mEAls With Less Salt：an Action to Reduce Salt Intake in School Meals for Children in Rural China
Acronym: HEALS-child
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Collaborators: China development research foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023157
Record Dates: First submitted 2023-10-09; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-09

CONDITIONS: Blood Pressure
Keywords: Salt reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Main study intervention- Salt substitute (Experimental): Replacing usual salt with salt substitute in school meals
  Interventions: Other: Main study intervention-Salt substitute
- Main study control- Usual salt (Placebo Comparator): Using usual salt in school meals
  Interventions: Other: Main study control-Usual salt
- Ancillary study intervention- Meal tray (Experimental): Replacing bowls with trays in school cafeteria
  Interventions: Other: Ancillary study intervention-Meal trays
- Ancillary study control- Bowl (Placebo Comparator): Using bowls in school cafeteria
  Interventions: Other: Ancillary study control-Bowls

INTERVENTIONS:
Other: Main study intervention-Salt substitute — replacing regular salt with salt substitute in school meals
  Arms: Main study intervention- Salt substitute
Other: Main study control-Usual salt — Use usual salt in school meals
  Arms: Main study control- Usual salt
Other: Ancillary study intervention-Meal trays — Replacing bowls with trays in school cafeteria
  Arms: Ancillary study intervention- Meal tray
Other: Ancillary study control-Bowls — Use bowls in school cafeteria
  Arms: Ancillary study control- Bowl

SUMMARY:
This study aims to assess the impact of the HEALS-Child action project on children's health in rural China. The goal of the project is to evaluate the effectiveness, feasibility, safety and cost-effectiveness of two salt reduction strategies: replacing usual salt with salt substitute in school meals, and replacing bowls with trays in school cafeteria. The study has two parts: the main study evaluates the salt substitute intervention, and the ancillary study evaluates the tray intervention. In the main study, over 16000 students from around 320 elementary or junior high school in rural China will be cluster-randomized into the two groups: 1. Salt substitute 2.usual salt. The primary outcome in the main study will be the change in systolic blood pressure. In the ancillary study, over 500 students from 10 elementary or junior high school will be cluster-randomized into the two groups: 1. meal trays 2.bowls. The primary outcome in the ancillary study will be the change in spot urine sodium. The interventions will last over 1 years. To evaluate the impact of interventions, 50 students were randomly selected from each school.

DETAILED DESCRIPTION:
The HEALS-Child action（Healthy School mEAls With Less Salt：an Action to Reduce Salt Intake in School Meals for Children in Rural China）is a project launched by China Development Research Foundation, aiming to reduce the salt in school meals and improve the nutrition for rural students. The goal of the study is to evaluate the effectiveness, feasibility, safety and cost-effectiveness of two salt reduction strategies: replacing usual salt with salt substitute in school meals, and replacing bowls with trays in school cafeteria. The study has two parts: the main study evaluates the salt substitute intervention, and the ancillary study evaluates the tray intervention.

1. Main study:

1. Aims:

   The aim in the main study is to test if replacing usual salt with the market available salt substitute in school meals could significantly reduce systolic blood pressure among rural school student. The corresponding null hypotheses in the main study is: the mean change from the baseline in systolic blood pressure of the students in schools that are supplied with salt substitute is equal to that in schools that are supplied with usual salt.
2. Study design:

   In the main study, over 16000 students from around 320 elementary or junior high school in rural China will be cluster-randomized into the two groups: 1. Salt substitute 2.usual salt. The salt substitute (NaCl 75% and KCl 25%) will be centrally provided. The intervention will last for two semesters(around 10-months).

   Before starting the intervention, 50 students were randomly selected from each school, and blood pressure, spot urine sodium and potassium and other indicators were measured at baseline.

   The randomization will be conducted centrally by the study coordinating center at Peking University Clinical Research Institute, after the baseline survey completed.

   The students will be followed up for blood pressure measurements and urine collection at the end of the first and second semesters after the intervention.
3. Outcomes:

   The primary outcome in the main study is the change in systolic blood pressure from baseline to follow-up. The secondary outcomes in the main study includes: The incidence of hypertension, the change in DBP, spot urine potassium, spot urine sodium, incremental cost-effectiveness ratio (ICER).
4. Power analysis and statistical analysis:

   On the assumptions of an intraclass correlation of 0.02, the number of clusters of 320 and 50 students in each school, and an α value of 0.05, the study to detect a mean 0.8 mmHg reduction in systolic blood pressure (SD, 10 mm Hg) between the intervention groups would have a power of 94.8%.

   Linear models adjusted for clustering based on participants with available measures were used to assess continuous outcomes. Generalized linear mixed model were used for analysis of effects on categorical outcomes.
5. Ethical considerations:

The study will be submitted to and approved by the Peking University IRB, which has the full accreditation from AAHRRP. The study salt substitute is the product available on Chinese market and has been approved manufactured according to the product standards issued by the ministry of health.

2. Ancillary study:

1. Aims:

   The aim in the ancillary study is to test if replacing bowls with trays in school cafeteria could significantly reduce spot urine sodium among rural school student. The corresponding null hypotheses in the ancillary study is: the mean change from the baseline in spot urine sodium of the students in schools that are supplied with meal trays is equal to that in schools that using bowls.
2. Study design:

   In the ancillary study, around 500 students from 10 elementary or junior high school in rural China will be cluster-randomized into the two groups: 1. meal trays 2.bowls. The meal trays will be centrally provided. The intervention will last for two semesters (around 10-months).

   Before starting the intervention, 50 students were randomly selected from each school, spot urine sodium and other indicators were measured at baseline.

   The randomization will be conducted centrally by the study coordinating center at Peking University Clinical Research Institute, after the baseline survey completed.

   The students will be followed up for urine collection at the end of the first and second semesters after the intervention.
3. Outcomes:

   The primary outcome in the ancillary study is the change in spot urine sodium from baseline to follow-up. The secondary outcomes in the ancillary study includes incremental cost-effectiveness ratio (ICER).
4. Power analysis and statistical analysis:

   On the assumptions of an intraclass correlation of 0.02, the number of clusters of 10 and 50 students in each school, and an α value of 0.05, the study to detect a mean 1g reduction in spot urine sodium (SD, 2.15g) between the intervention groups would have a power of 90.0%.

   Linear models adjusted for clustering based on participants with available measures were used to assess continuous outcomes.
5. Ethical considerations:

The study will be submitted to and approved by the Peking University IRB, which has the full accreditation from AAHRRP.

ELIGIBILITY:
Inclusion criteria:

Attend school stably in this academic year, and expect to take no more than one month of leave for the whole academic year； Have lunch at school at least three times a week.

Exclusion criteria:

Unable to complete the baseline blood pressure measurement and spot urine collection.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16000 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Primary outcome for the main study-Systolic blood pressure | 10-month
  The change in systolic blood pressure from baseline to follow-up
Primary outcome for the ancillary study-Spot urinary sodium | 10-month
  The change in spot urinary sodium from baseline to follow-up

SECONDARY OUTCOMES:
Secondary outcome for the main study-Incidence of hypertension | 10-month
  The new-onset hypertension during study period
Secondary outcome for the main study-Spot urinary sodium | 10-month
  The change in spot urinary sodium from baseline to follow-up
Secondary outcome for the main study-Spot urinary potassium | 10-month
  The change in spot urinary potassium from baseline to follow-up
Secondary outcome for the main study-Diastolic blood pressure | 10-month
  The change in diastolic blood pressure from baseline to follow-up
Secondary outcome for the main study-ICER | 10-month
  Incremental cost-effectiveness ratio, defined by the difference in the cost for every unit of gain in the pertained effectiveness outcome
Secondary outcome for the ancillary study-ICER | 10-month
  Incremental cost-effectiveness ratio, defined by the difference in the cost for every unit of gain in the pertained effectiveness outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yangfeng Wu, PhD, Principal Investigator — Peking University

IPD SHARING:
Plan to Share IPD: No